CLINICAL TRIAL: NCT00851032
Title: An Initiative for Molecular Profiling in Advanced Cancer Therapy (IMPACT) Trial. A Molecular Profile-Based Study in Patients With Advanced Cancer Treated in the Investigational Cancer Therapeutics Program
Brief Title: Initiative for Molecular Profiling in Advanced Cancer Therapy (IMPACT) Trial, An Umbrella Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2007-0885; 1UL1RR024148 (NIH)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancer; Initiative for Molecular Profiling in Advanced Cancer Therapy; IMPACT; Molecular Profile-Based Study; Investigational Cancer Therapeutics Program; Molecular profiling; Phase I Therapies; Tissue Bank
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Specimen obtained from MDACC Tissue Bank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Molecular Profiling Analyses: Participants seen in the Department of Investigational Cancer Therapeutics at MD Anderson Cancer Center in Houston, Texas
  Interventions: Other: Molecular Profiling Analyses

INTERVENTIONS:
Other: Molecular Profiling Analyses — Molecular profiling analyses from advanced cancer participants' stored tissue bank samples.

SUMMARY:
Primary Objective The primary objective of this study is to establish a program for the molecular profiling of patients with advanced cancer, with the goals of (1) providing a comprehensive characterization of the molecular profiles of individual patients and (2) correlating molecular profile with response to phase I therapies.

Specimens will be received from the LAB07-0817 (Tissue Bank) protocol in the Department of Investigational Cancer Therapeutics. Note that this study is considered an umbrella protocol to systematically enroll phase I patients for molecular profiling analysis and correlate the results with treatment outcomes. The IMPACT trial is not a treatment protocol.

Secondary Objectives

1. To characterize advanced cancer by delineating genetic mutations, amplifications, translocations, and other defining molecular patient characteristics.
2. To assess the antitumor effects of treatments by tumor responses using the World Health Organization (WHO) or Response Evaluation Criteria in Solid Tumors (RECIST) criteria and/or any other clinical benefits, including progression-free survival and overall survival, demonstrated in phase I clinical trials.
3. To correlate molecular profiles of patients with evidence of antitumor activity (complete remission, partial remission, prolonged stable disease, or overall survival) to define subsets of patients who will respond to specific therapies in clinical trials of novel agents.
4. To correlate molecular profiles with toxicities induced by investigational agents to define subsets of patients who may or may not be candidates for treatment with these agents in the future.

DETAILED DESCRIPTION:
The prognosis of patients with advanced metastatic malignancies is poor, and their median survival, irrespective of diagnosis, is approximately 8.8 months (95% confidence interval, 7.4 to 10.9 months). In recent years there has been increased interest in novel agents.

Elucidating the molecular basis of advanced cancer will lead to the development of potentially curative strategies for these diseases aimed at the specific molecular and genetic aberrations characteristic of specific tumors.

This study is a molecular profiling analyses of the patients' stored samples and will not involve more than minimal risk to the subjects. Subjects are at no more than minimal risk because only leftover blood, tissue, and patient data will be used for this study, and all patient data will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

1) Any patient seen in the department of Investigational Cancer Therapeutics is eligible. Patients who have blood or tissue samples collected must be registered on the tissue bank protocol (LAB07-0817).

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Advanced Cancer Treated in the Investigational Cancer Therapeutics Program Registered on MDACC tissue bank protocol (LAB07-0817).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-02 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Establish a program for the molecular profiling of patients with advanced cancer. | 6 Years
  For characterizing the molecular profile, descriptive statistics and exploratory data analysis performed first. Categorical data described using contingency tables. Continuously scaled measures summarized with descriptive statistical measures (i.e., mean (± s.d.) and median (range)). Distribution plots such as histograms and box plots applied.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Tsimberidou AM, Hong DS, Wheler JJ, Falchook GS, Janku F, Naing A, Fu S, Piha-Paul S, Cartwright C, Broaddus RR, Nogueras Gonzalez GM, Hwu P, Kurzrock R. Long-term overall survival and prognostic score predicting survival: the IMPACT study in precision medicine. J Hematol Oncol. 2019 Dec 30;12(1):145. doi: 10.1186/s13045-019-0835-1. PMID 31888672
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org